CLINICAL TRIAL: NCT03740854
Title: The Effects of Two Different Ventilation Strategies on Lung Ventilation in Patients Undergoing Robotic Radical Prostatectomy: Ultrasonographic Evaluation.
Brief Title: The Effects of Two Different Ventilation Strategies on Lung Ventilation: An Ultrasonographic Evaluation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Hacer Zeynep Turgut, MD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 68839
Record Dates: First submitted 2018-11-12; First posted 2018-11-14 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: lung ultrasonography; mechanical ventilation; pressure controlled ventilation; volume controlled ventilation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure Controlled Ventilation (Active Comparator): Patients undergoing pressure controlled ventilation
  Interventions: Other: Pressure Controlled Ventilation
- Volume Controlled Ventilation (Active Comparator): Patients undergoing volume controlled ventilation
  Interventions: Other: Volume Controlled Ventilation

INTERVENTIONS:
Other: Pressure Controlled Ventilation — Patients will be ventilated with a pressure level which supplies a tidal volume corresponding 8ml/kg, 12 breaths per minute, 1/2 inspiration/expiration ratio and %40 Fraction of Inspired Oxygen . These ventilator settings can be changed in order to adjust end tidal carbon dioxide and oxygen saturation levels.
  Arms: Pressure Controlled Ventilation
Other: Volume Controlled Ventilation — Patients will be ventilated with a tidal volume which corresponds 8ml/kg, 12 breaths per minute, 1/2 inspirastion/expiration ratio and %40 Fraction of Inspired Oxygen . These ventilator settings can be changed in order to adjust end tidal carbon dioxide and oxygen saturation levels.
  Arms: Volume Controlled Ventilation

SUMMARY:
This study will be performed in robotic assisted laparoscopic radical prostatectomy patients in Cerrahpasa Medical Faculty Monoblock Operating Room. Since robot-assisted laparoscopic radical prostatectomy is a surgical procedure which requires long-term mechanical ventilation, excessive trendelenburg position (30-45 °) and pneumoperitoneum; these interventions may lead to respiratory complications such as ventilation difficulty and aeration loss in patients. Nowadays, lung ultrasonography has been used in anesthesia practice and intensive care units in order to determine lung aeration loss. In this study, the investigators aimed to compare the possible aeration loss in lung parenchyma during pressure controlled ventilation and volume controlled ventilation which are frequently used in anesthesia practice in patients undergoing robotic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria: 18-75 age

* Patient who will be undergo robot assisted laparoscopic prostatectomy surgery
* Patient with ASA (American Society of Anesthesiologists) Score 1-3

Exclusion Criteria:

* Patients with ASA Score above 3
* Patients with obstructive (FEV1<%60) or restrictive pulmonary disease (FVC<%60)
* Patients with intrathoracic operation history
* Heavy smokers (>25 cigarettes/day)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since our study will be performed in patients with prostate cancer, all of our patients will be male.
Enrollment: 72 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
The difference between LUS Scores at T5 in patients ventilated with VCV and PCV | (T5) 60 minutes after patients come to the recovery room.
  Lung Ultrasonography will be applied to patients after surgery in the recovery room at T5. Two different groups' LUS scores will be calculated and compared.

SECONDARY OUTCOMES:
The difference between LUS Scores at T2 in patients ventilated with VCV and PCV | (T2) 5 minutes after intubation
  Lung Ultrasonography will be applied to patients after intubation. Two different groups' LUS scores will be calculated and compared.
The difference between LUS Scores at T3 in patients ventilated with VCV and PCV | (T3) 5 minutes after the surgical procedure is finished
  Lung Ultrasonography will be applied to patients at Trendelenburg position after the surgical prosedure is finished. Two different groups' LUS scores will be calculated and compared.
The difference between LUS Scores at T4 in patients ventilated with VCV and PCV | (T4) 5 minutes after taking the patient to supin position
  Lung Ultrasonography will be applied to patients at supin position after the surgical prosedure is finished. Two different groups' LUS scores will be calculated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Fatis Altintas, MD, Study Director — Istanbul Unıversity-Cerrahpasa, Cerrahpasa Medical Faculty
Locations (1):
- Medical Faculty of Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided